CLINICAL TRIAL: NCT01228500
Title: The Use of Bioscaffolds in Conjunction With Negative Pressure Therapy: A Prospective Randomized Double-Blinded Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TEI-001
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Arm (Internal Control) (Experimental): One-half of ulcer receives negative pressure wound therapy
  One-half of ulcer receives a fetal bovine collagen bioscaffold (PriMatrix, TEI Biosciences, Boston, MA) in addition to the same negative pressure wound therapy
  Interventions: Device: PriMatrix

INTERVENTIONS:
Device: PriMatrix — Dermal Repair Scaffold

SUMMARY:
The primary aim of this study proposal is to test an innovative form of fetal bovine dermis bioscaffold in combination with negative pressure wound therapy (NPWT) to enhance wound healing in diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Adult Type 1 or 2 diabetic patients that present with foot ulcers.
* Ulcer size of at least 3 centimeters (cm) in diameter at its widest dimension.
* Ulcer depth: Full thickness (absence of all epithelial layers or deeper)
* Adequate perfusion (at least one palpable pedal pulse or pedal bypass graft)
* All ulcer durations will be eligible
* Patients currently receiving NPWT for a diabetic foot ulcer
* Patients must be appropriate NPWT candidates and be willing and able to sleep, ambulate, and rest with the NPWT unit in place.

Exclusion Criteria:

* Active foot infections
* Presence of any serious disease including end-stage renal failure requiring dialysis or renal transplantation or active malignant disease requiring treatment which seriously compromises the patient's ability to complete this study
* Patients who are pregnant
* Allergies to any material contained within the NPWT or bioscaffold
* Any condition that would exclude NPWT use including but not limited to active bleeding, presence of malignancy in the wound or inability to follow any of the NPWT safety guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Time to healing | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Cook, DPM, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States